CLINICAL TRIAL: NCT01885377
Title: SWESS: The SWedish Exercise Shoulder Study in Primary Care for Patients With Subacromial Pain - a Randomized Clinical Trial
Brief Title: SWESS: The SWedish Exercise Shoulder Study in Primary Care for Patients With Subacromial Pain
Acronym: SWESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Collaborators: University Hospital, Linkoeping (Other); Ostergotland County Council, Sweden (Other)
Responsible Party: Principal Investigator, Kajsa Johansson, Senior Lecturer, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 8820 PV-JN-1
Record Dates: First submitted 2013-06-18; First posted 2013-06-25 (Estimated); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Shoulder Pain; Shoulder Impingement Syndrome; Disorder of Rotator Cuff; Subacromial Bursitis
Keywords: Subacromial pain; Impingement; Exercises; Physical therapy; Primary care
MeSH Terms: conditions — Shoulder Pain; Shoulder Impingement Syndrome; Motor Activity | interventions — Posture; Exercise Movement Techniques

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Specific exercise group (Experimental): A progressive program of strength-endurance exercises for the rotator cuff and scapula stabilizing muscles combined with mobilization of the joint capsule when needed
  Interventions: Other: Specific exercise group
- Control exercise group (Active Comparator): General movements for the neck and shoulder and self-stretching. No progression some addition of exercises during the three month period.
  Interventions: Other: Control exercise group

INTERVENTIONS:
Other: Specific exercise group — A program where exercise load is individually adjusted and the exercises progressed during a 3 month period. The 'pain monitoring model' were used to find the individual resistance. Several exercises are performed eccentrically in order to load more. Initially the exercises were PT-tutored every week and then every other week.
  Other Names: •Strength-endurance exercises; •Rotator cuff; •Scapular stabilization; •Eccentric; •Posture
  Arms: Specific exercise group
Other: Control exercise group — A program with movements to maintain flexibility in the neck and shoulder muscles. Initially PT-tutored every week and then every other week.
  Other Names: •Movement exercises; •Stretching; •Posture
  Arms: Control exercise group

SUMMARY:
Objective: A randomized clinical trial in order to evaluate the efficacy of a specific exercise strategy for patients with subacromial pain.

Hypothesis:

H1 - The three month specific exercise strategy has a satisfactory effect improving shoulder function and/or shoulder pain.

H0 - No difference between the two exercise strategies (specific exercise strategy and active control exercises).

Method: Patients attending primary care with subacromial pain are offered participation. If accepted, they will participate in a three month rehabilitation program. The duration of symptoms can vary from 2 weeks and longer. The patients will be randomized to either rehabilitation; the specific exercise strategy or active control exercises. All patients has an equal number of sessions with the physical therapist (PT) to offer similar attention and support with exercise performance. A blinded physical therapist evaluates the following outcomes at baseline and after three-, six and twelve months:

Primary outcomes: Constant-Murley shoulder assessment (CM-score). Secondary outcomes; Disabilities of the Arm Shoulder and Hand questionnaire (DASH), different aspects of pain by Visual Analogue Scale (VAS), EuroQol-5D index (EQ-5D) and EuroQol-VAS (EQ-VAS), The Patient Specific functional Scale, and Patients' global impression of change (PGIC). Also sick-leave and return to work will be recorded. All patients are evaluated with a diagnostic ultrasound to reveal the status of the rotator cuff.

Additional to the analysis of treatment effect on shoulder function and pain, factors influencing and explaining the CM-score at follow-ups will be analyzed.

This study is warranted in order to evaluate if an earlier reported positive effect on shoulder function and pain with the specific exercise strategy, in patients on waiting list for subacromial decompression, can be repeated in the primary care population of patients with subacromial pain. There is no consensus about first-line exercises for patients with subacromial pain, and these positive results on pain and shoulder function need to be reproduced in primary care before they can be recommended and implemented. Further, knowledge about which factors that can be used in prediction rules for patients that will respond to the exercises or needs surgery is lacking.

DETAILED DESCRIPTION:
This study will be reopened and will continue the inclusion due to underpowered results.

A new application to the Ethical committee was submitted. Approval to reopen this RCT-study was received at 27th of September 2018 (dnr 218/445-32).

Additional inclusion of 40 additional patients will start at 1th of November 2018. Data from baseline to 12 months follow-up (as described in protocol) will be collected. Inclusion continued and the last inklusion was completed in February 2020. Data Collection for all follow ups is anticipated to be completed at latest during March the year of 2021.

ELIGIBILITY:
Inclusion Criteria:

* At least 2 weeks of symptom duration
* Typical history and pain location (C5 dermatome)

Three of these four must be positive:

* Neer impingement sign
* Hawkins-Kennedy impingement sign
* Jobe supraspinatus test
* Patte maneuver

Exclusion Criteria:

* Polyarthritis or fibromyalgia
* Pathological hyper-laxity or dislocation of the any of the shoulder joints
* Cervical spine pathology
* Lack of communication skills that prevent the use of outcome measures
* Signs in ultrasound of bone spurs i.e. Acromio-Clavicular joint, that will affect the subacromial space

Ages: 30 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2020-03 (Actual); Study Completion 2021-03 (Actual)

PRIMARY OUTCOMES:
The Constant-Murley shoulder assessment | Baseline and change 3-, 6- and 12 months
  Measure a combination of self assessed and clinician assessed items; pain, range-of-motion (flexion and abduction), functional positions (hand in neck as well as hand in back), abduction strength.
  The score is summarized to a maximum of 100 for best available shoulder function.

SECONDARY OUTCOMES:
Euro Qol 5D index (EQ 5D) | Baseline and change 3-, 6- and 12 months
  Health Related Quality of Life by EuroQol 5 dimensions and index. Measures different items related to heath related quality of life: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. It results in a health-state where an index of 1 is optimal.
Disabilities of the arm, shoulder and hand | Baseline and change 3-, 6- and 12 months
  Self-assessment of the ability to performed exemplified activities. 0 indicates a non-affected upper extremity.
VAS for pain | Baseline and change 3-, 6- and 12 months
  Self-assessed for pain at rest, in activity and at night if it disturbs sleeping
Patients Global Impression of Change (PGIC) | At follow-up: 3-, 6- and 12 months
  The patients are asked to assess change. A scale ranging from getting worse by the intervention to be recovered.
The Patient Specific functional Scale | Baseline and change 3-, 6- and 12 months
  Self-selected functional activities to relate efficacy to during follow-ups.
Euro Qol VAS (EQ VAS) | Baseline and change 3-, 6- and 12 months
  In EQ VAS the patients assess their health state on a vertical line valued from 0-100.

OTHER OUTCOMES:
Hospital Anxiety and Depression Scale (HAD) | Baseline
  To screen mental health (depression and/or anxiety) in all included patients. Maximum score is 21 points for the depression and anxiety part respectively. The higher score, the higher risk of a depression and/or anxiety.
Sick-leave and return to work or working status | Baseline, 3-, 6- and 12 months
  Patient reported can be double checked by the Swedish Social Insurance Agency.

CONTACTS AND LOCATIONS:
Overall Officials: Birgitta Öberg, Professor, Study Chair — Div. of Physical Therapy, Dept. of Medical and Health Sciences, Linköping University; Lars Adolfsson, Professor, Study Director — Dept. of Orthopaedics, University Hospital Linköping & Linköping University; Kajsa Johansson, PhD, Principal Investigator — Div. of Physical Therapy, Dept. of Medical and Health Sciences, Linköping University
Locations (1):
- Primary Care unit "Rörelse & Hälsa", Linköping, Sweden

REFERENCES:
- [Background] PMID: 22349588